CLINICAL TRIAL: NCT00384592
Title: A Study to Assess the Effectiveness of Esomeprazole 40 mg Once Daily in Subjects With Continuing Gastroesophageal Reflux Disease (GORD) Symptoms Following Treatment Wit a Previous Full Dose Proton Pump Inhibitor (PPI)
Brief Title: PPI Sequencing Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00104
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Gastro-Oesophageal Reflux Disease
Keywords: heartburn; reflux; proton pump inhibitor; GERD; GORD
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole; Restraint, Physical

INTERVENTIONS:
Drug: Esomeprazole
Procedure: Physical exam
Procedure: Pregnancy test if applicable

SUMMARY:
The purpose of this study is to assess how patients with gastro-oesophageal reflux disease (heartburn) who are currently receiving treatment with a proton pump inhibitor but are still experiencing symptoms will benefit from a change in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persisting symptoms of GORD despite previous treatment with a full dose proton pump inhibitor
* Informed consent
* Over 18 years of age

Exclusion Criteria:

* Current course of Proton Pump inhibitor treatment for more than 8 weeks prior to enrolment in the study;
* More than 1 other course of PPI treatment in the previous 12 month;
* Previous use of esomeprazole;
* Presence of alarm symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the change in the frequency of heartburn from baseline value at entry to the end of the study, after 8-weeks treatment with esomeprazole 40mg compared to previous full dose treatment with a PPI daily

SECONDARY OUTCOMES:
Change in frequency and severity of heartburn, epigastric pain and acid regurgitation after 4 and 8 weeks treatment from baseline value at study entry
Change in symptom control from baseline to 4 and 8 weeks using QOL questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Rhiannon Rowsell, MD, Study Director — AstraZeneca; Roger Jones, MD, Principal Investigator — UCL
Locations (14):
- United Kingdom (14):
  - Research Site, Allerton
  - Research Site, Ashford
  - Research Site, Atherstone
  - Research Site, Ayrshire
  - Research Site, Bath
  - Research Site, Blackpool
  - Research SIte, Bolton
  - Research Site, Coventry
  - Research Site, Fowey
  - Research SIte, Glasgow
  - Research Site, Hamilton
  - Research Site, Motherwell
  - Research Site, Stevenage
  - Research Site, Warminster